CLINICAL TRIAL: NCT01583946
Title: Temporally-Oriented Subjective Well-being Across Transitions-Resources & Outcomes
Acronym: LIFT
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Rachel Hess, MD, University of Pittsburgh
Other Study IDs: PRO11070243; 1R01AT007262-01 (NIH)
Record Dates: First submitted 2012-04-17; First posted 2012-04-24 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2015-12

CONDITIONS: Quality of Life
Keywords: subjective well-being; life transitions; health-related quality of life; health; healthcare costs

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Male low past-oriented SWB
- Male high past-oriented SWB
- Female low past-oriented SWB
- Female high past-oriented SWB
- Black Female high past-oriented SWB
- Black Female low past-oriented SWB
- Black male low past-oriented SWB
- Black male high past-oriented SWB

SUMMARY:
As individuals age, they undergo transitions in many aspects of their lives. These transitions include social, economic and health transitions. People review their lives, and reflect on past choices. Future time is limited by the increasing proximity to end of life. This may lead to regrets and, in people with the ability to use compensatory mechanisms, a redoubling of efforts to achieve valued goals or a reprioritization of valued goals. In the context of aging, individuals' past, present, and future-oriented subjective well-being (SWB) may change. There is an incomplete understanding of the relationship of SWB, intra- and inter-personal resources, and outcomes, (particularly health and healthcare-cost outcomes). These issues have complicated the use of SWB measures and the investigators are left with traditional metrics such as life expectancy, infant mortality, wealth, and poverty to assess healthy aging, resulting in an incomplete picture of healthy aging. This project will examine the relationships among SWB, intra- and inter-personal resources, and health and healthcare-cost outcomes. It will advance the understanding of SWB and its role in healthy aging in order to assist policy makers in valuing the potential benefits of improving SWB on health and healthcare costs. The investigators will accomplish this through the following specific aim:

Aim 1: To determine how SWB (past, present, and future-oriented): (1) is affected by life transitions, and (2) affects outcomes after life transitions.

DETAILED DESCRIPTION:
Aim: To determine how Subjective Well-Being (SWB; past, present, and future-oriented): (1) is affected by life transitions, and (2) affects outcomes after life transitions.

Rationale: Social, economic, and health transitions are common in aging populations. Adaptation to these transitions likely impacts SWB and therefore may alter subsequent health and healthcare-cost outcomes.

Hypotheses: Negative life transitions will negatively impact assessments of present and future-oriented SWB and result in worse health and healthcare-cost outcomes. More positive intra- and inter-personal resources will lessen this impact. Having better present or future-oriented SWB will diminish the impact of the transition on health and healthcare-cost outcomes.

Approach: Investigators will establish an observational cohort of adults aged 50 and older (n=600) seen in the same primary care practice stratified by gender, race, and SWB. Investigators will collect information at baseline and each of two annual follow-up assessments regarding SWB, intra- and inter-personal resources, and outcomes. Investigators will compare those who experience life transitions to those who do not in terms of their changes in the temporal perspectives of SWB, health, and healthcare-cost outcomes.

The successful completion of this project will disentangle temporal perspectives in SWB, further the understanding of the impact of aging and life transitions on SWB, relate individuals' SWB to health and healthcare-cost outcomes, and clarify the relationship of experienced SWB to evaluative SWB, all within the context of intra- and inter-personal resources. It will enable researchers, clinicians, and policy makers to better use SWB as a metric assessing the health and welfare of individuals and societies. The study population is primarily older adults from a primary care practice, University of Pittsburgh's General Internal Medicine Oakland (GIMO).

Aim: To determine how SWB (past, present, and future-oriented): 1) is affected by life transitions and 2) affects outcomes after life transitions.

C.2.a. Overview of the Aim Social, economic, and health transitions, commonly occur in aging populations. Adaptation to these transitions likely impacts SWB and subsequent health and healthcare-cost outcomes.

Investigators will enroll a purposive sample (n=600) of adults aged 50 and older seen at the GIMO primary care practice. Investigators will collect information at baseline and each of two annual follow-up assessments regarding SWB, intra- and inter-personal resources and outcomes. Investigators will compare those who experience life transitions to those who do not in terms of their changes in temporally-oriented SWB and health and healthcare-cost outcomes.

Measures In addition to basic demographics including age, gender, ethnicity, race, educational attainment, marital status, and employment status, investigators will collect data described below.

Subjective Well-Being. Investigators will use the temporal measure of SWB by Pavot, Deiner, and Suh8 which includes 15 items-5 representing each of past, present, and future-oriented SWB.

Intra- and inter-personal resources. These constructs were selected because they are important to the understanding of SWB and the relationships between SWB and the outcomes tested in our model. Each instrument has been related to health outcomes, healthcare-cost outcomes, SWB, and/or health-related quality of life in prior work and key citations are provided. Bringing together such a comprehensive assessment battery to understand temporally-oriented SWB and its relationship to these measures and outcomes, the impact of transitions on these relationships, and the relationship of experiences and experienced SWB to evaluative SWB, as proposed in the current project, is necessary to advance the field.

Definition of transitions. Separate groups will be defined for those who undergo, or do not undergo, three broad categories of transitions: social, economic, and health, or any of the three transitions; individuals may have more than one type transition. In addition to "any" transition, each transition type will be analyzed separately. As described in the significance section, investigators have found that these transitions are common in older adults. Participants will complete items from the Life Events Scale at each time-point. Investigators will use MARS and EpicCare to identify any new health conditions (based on additions to the problem list or past medical history) supplement the identification of health transitions.

Health and healthcare costs. Investigators will use health and healthcare costs to assess the predictive validity of our measure in the Primary care sample. Health and healthcare-cost measures will be obtained from both the using the Medical Archival System (MARS)43 and the EpicCare electronic medical record (EMR). MARS data include all patients seen at the University of Pittsburgh Medical Center's (UPMC) twenty hospitals, four long-term care facilities, and 350 physician offices and outpatient clinics. The MARS repository houses 209 million clinical reports, 460 million financial transactions, and patient demographic information. EpicCare, GIMO's EMR, electronically contains all information required in a traditional paper medical record. All documentation (including past medical history), orders, and results are captured. Any paper result, for example laboratory testing done out of state, is abstracted as discrete data items into EpicCare. The primary measure will be healthcare costs. Cost outcomes, from MARS and EpicCare, will include the total healthcare charges documented within the UPMC system (including outpatient prescription medications at the average retail cost) in the year following the assessment. As the largest provider of care in Western Pennsylvania, UPMC delivers the vast majority of care received by GIMO patients.

Why use costs as the primary measure in this sample? Healthcare costs provide a relatively simple summary of overall care intensity across people with a variety of health concerns and is particularly relevant to health policy. It is broadly applicable and is responsive to this request for applications. Two alternative endpoints are diagnosis of a new medical condition or disease management process measures. Based on our prior experience, we expect the majority of participants to develop new medical conditions, so treating a new diagnosis as the primary measure would give minimal variation in the measure and would limit our ability to see a difference based on temporally associated SWB. GIMO's clinical variety makes disease management process measures an impractical primary measure. Investigators have chosen to examine two common primary care conditions, diabetes and coronary artery disease, that require both patient and physician participation in management as a secondary measure.

Secondary health measures will include (1) number of new diagnoses developed, (2) hospitalization (yes or no) and, among those hospitalized, length of stay, and (3) disease management over one year. Investigators will track the development of the following conditions identified by Verbrugge and Patrick: arthritis, visual impairment, hearing impairment, ischemic heart disease, hypertension, chronic obstructive pulmonary disease, diabetes mellitus, and malignant neoplasm.42 A diagnosis will be considered new if it is used as a billing diagnosis and has not been used previously as a billing diagnosis or listed on the problem list or past medical history. Because all participants will have been seen in the past at GIMO we will be able to easily differentiate new from previously existing diagnoses. Hospitalization will be defined as admission to one of twenty UPMC medical or psychiatric hospitals and length of stay. Disease management will be based on percent of fulfilled quality metrics (total number of metrics fulfilled, divided by the total number of metrics) defined by NCQA44 and used as quality measures in GIMO.

ELIGIBILITY:
Inclusion Criteria:

* participants will be included if they are GIMO patients who complete the FAST,
* are aged 50 or older,
* agree to participate, and
* belong to an unfilled bin.

Exclusion Criteria:

* Investigators will exclude individuals from the purposive sample who do not provide informed consent. There will be no exclusion based on race, gender, immigration, or HIV status.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females 50 and older
Sampling Method: Non-Probability Sample
Enrollment: 793 (Actual)
Dates: Start 2012-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
healthcare costs | Over at least 3 years
  healthcare costs

SECONDARY OUTCOMES:
number of new diagnoses developed | Over at least 3 years
hospitalization | Over at least 3 years
  hospitalization (yes or no)
hospital length of stay | Over at least 3 years
  among those hospitalized, length of stay
disease management over one year | Over at least 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Hess, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- Division of General Internal Medicine UPMC Montefiore Hospital, Pittsburgh, Pennsylvania, United States